CLINICAL TRIAL: NCT03451578
Title: The Role of Alpha Melanocyte Stimulating Hormone in Ocular Disease
Brief Title: Alpha MSH in Ocular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00086021
Record Dates: First submitted 2018-02-26; First posted 2018-03-01 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Advanced Dry Macular Degeneration
Keywords: macular degeneration; blindness
MeSH Terms: conditions — Macular Degeneration; Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Advanced Dry macular degeneration (Other)
  Interventions: Device: Alpha MSH assay

INTERVENTIONS:
Device: Alpha MSH assay — Assay to detect levels of alpha MSH in intraocular fluid.

SUMMARY:
The purpose of this study is gain a better understanding of a molecule called alpha melanocyte stimulating hormone (alpha MSH) and its potential role in your retinal disease. Alpha MSH has been shown to have an important role in the regulation of ocular immunity in animal models of inflammatory retinal diseases and retinal dystrophies, and there may be a protective effect of alpha MSH. By studying the levels of alpha MSH in your eye we may better understand its role in advanced dry macular degeneration. By studying the levels of this molecule we hope to better understand if it may be a good target for future treatment.

DETAILED DESCRIPTION:
A small amount (0.1 mL) of aqueous humor would be removed from the study eye in the clinic setting. This sample will be processed and then sent off for measurement of alpha MSH levels.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* diagnosis of advanced dry macular degeneration with foveal geographic atrophy
* limited vision or blindness (20/100 or worse) in that eye
* pseudophakia (prior cataract surgery in that eye)

Exclusion Criteria:

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Fekrat, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Advanced Dry Macular Degeneration
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Advanced Dry Macular Degeneration
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Level of Alpha Melanocyte Stimulating Hormone as Measured by Enzyme-linked Immunosorbent Assay
Time Frame: 2 hours
Population: Unable to obtain alpha MSH levels.
Arm/Group | Advanced Dry Macular Degeneration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 visit, up to 2 hours
Arm/Group | Advanced Dry Macular Degeneration
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

LIMITATIONS AND CAVEATS:
The investigators found through various approaches that alpha MSH was not measurable within the samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT03451578/Prot_001.pdf